CLINICAL TRIAL: NCT02917681
Title: Study of Two Intrathecal Doses of Autologous Mesenchymal Stem Cells for Amyotrophic Lateral Sclerosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Pontifícia Universidade Católica do Paraná (Other)
Responsible Party: Principal Investigator, Gerson Chadi, Professor, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 401922/2014-6
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: AMYOTROPHIC LATERAL SCLEROSIS
Keywords: ALS; mesenchymal stem cells; intrathecal
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSC injection (Experimental): Patients will be followed for 3 months before bone marrow aspiration (BMA). Patients will receive 2 intrathecal MSC injections, 1 and 2 months after BMA. The patients will be followed for 6 months after the interventions.
  Interventions: Other: Two intrathecal MSC injections

INTERVENTIONS:
Other: Two intrathecal MSC injections

SUMMARY:
The study aims to evaluate primarily safety of two injections of autologous mesenchymal stem cells in Amyotrophic Lateral Sclerosis patients. Secondary outcomes of efficacy will also be evaluated

DETAILED DESCRIPTION:
The study is an open-label, unmasked, uncontrolled phase I and II trial to evaluate safety and efficacy of two injections of autologous mesenchymal stem cells (MSC) in Amyotrophic Lateral Sclerosis (ALS) patients. Patients will be recruited trough a web-based registration system, open for all ALS Brazilian patients. The patients will be enrolled after in-person screening at the University of Sao Paulo Medical School Clinics Hospital and inclusion criteria fulfilled. There will be 9 national calls for registration, two months apart each. The enrolled patients will be followed for 3 months before bone marrow aspiration (BMA). Patients will receive 2 intrathecal MSC injections, 1 and 2 months after BMA. The patients will be followed for 6 months after the interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70
2. Possible, probable or definite ALS following El Escorial Revised Criteria (Brooks, 2000)
3. ALSFRS-r ≥30 at enrollment
4. Forced Vital Capacity ≥65% of the height and weight standard
5. No-pregnancy agreement
6. Regional accessibility to the study site
7. Capability to give away agreed consensus
8. Patients will be followed at Academic Institutions at their hometown

Exclusion Criteria:

1. Previous cellular therapy
2. Incapacity to lay still during bone marrow aspirate or intrathecal MSC injections
3. Personal history of auto-Immune, myeloproliferative or myelodysplastic diseases, leukemia, lymphoma, whole-body irradiation, hip fracture, severe scoliosis or incapacity to undergo any of the study's proposed procedures
4. Any other disease that may interfere with the study
5. Any other neurological diseases
6. Aspartate or alanine aminotransferases elevated >3x normality upper limit
7. Serum creatinine >2x normality upper limit
8. Hepatitis B and C, HIV, HTLV I and II and syphilis
9. Immunosuppressant drug use within 6 weeks from the study's screening
10. Pregnancy or breast-feeding
11. Acquired or inherited Immunodeficiency
12. Participation in other clinical trials
13. Non-invasive ventilation, tracheostomy or diaphragm pacing
14. Substance abuse within one year and other unstable mental health diseases according to researcher's judgement
15. Gastrostomy or any alternative feeding means
16. Inappropriate in-vitro MSC expansion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-02 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Safety | 10 months
  Clinical and laboratory monitoring of possible reactions to intrathecal MSC delivery

SECONDARY OUTCOMES:
Change in Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) | 10 months
  Specific scale for assessing ALS disease progression
Change in Handheld dynamometry | 10 months
Change in Electrical Impedance Myography | 10 months
Change in Forced Vital Capacity (FVC) | 10 months
Change in Isometric Strength | 10 months
Changes in morphometric parameters of MRI of encephalon and spinal cord | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerson Chadi, MD, PhD, Principal Investigator — Full Professor
Locations (1):
- University of Sao Paulo School of Medicine Clinics Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No